CLINICAL TRIAL: NCT04898959
Title: Psychometric Evaluation of the Arabic Activity-specific Balance Confidence (A-ABC) and the Arabic Prosthetic Mobility Questionnaire (PMQ) in Saudi Lower Amputees
Brief Title: Psychometric Evaluation of the Arabic Activity-specific Balance Confidence (A-ABC) and the Arabic Prosthetic Mobility Questionnaire (PMQ)
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2021.575
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-05

CONDITIONS: Filling Out Questionnaires
Keywords: Arabic Activity-specific Balance Confidence; Arabic Prosthetic Mobility Questionnaire; Psychometric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Lower extremity amputees
  Interventions: Other: Filling out Questionaire

INTERVENTIONS:
Other: Filling out Questionaire — Filling out the Arabic Activity Specific Balance Confidence (A-ABC) and the Arabic Prosthetic Mobility Questionnaire twice at 2-3 week intervals

SUMMARY:
The primary aim of this study is to perform perform a psychometric analysis of Arabic Activity-specific Balance Confidence (A-ABC) and the Arabic Prosthetic Mobility Questionnaire (A-PMQ) through a modern psychometric approach involving Rasch analysis (RA) to enable its use among Arabic speaking population and to enhance confidence in its use patients with lower limb amputation.

ELIGIBILITY:
Inclusion Criteria:

* current users of lower limb prosthesis of minum 6 month,
* to be able to fully understand and appropriately complete the questionnaire,
* to be unilater amputee.

Exclusion Criteria:

* inability to understand and complete the questionnair (e.g. cognitive or language impairment; not native-Arabic speaker),
* less the 6 month of using the prosthesis,
* bilateral and partial lower limb amputees

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Unilateral lower limb amputees (above ankle dezarticulation level)
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Rasch analysis | Change from baseline answers of questions following 3 weeks
  to perform a psychometric analysis of Arabic Activity-specific Balance Confidence (A-ABC) and the Arabic Prosthetic Mobility Questionnaire (A-PMQ) through a modern psychometric approach involving Rasch analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Franchignoni F, Monticone M, Giordano A, Rocca B. Rasch validation of the Prosthetic Mobility Questionnaire: A new outcome measure for assessing mobility in people with lower limb amputation. J Rehabil Med. 2015 May;47(5):460-5. doi: 10.2340/16501977-1954. PMID 25783231
- [Result] Alghwiri AA, Alghadir AH, Al-Momani MO, Whitney SL. The activities-specific balance confidence scale and berg balance scale: Reliability and validity in Arabic-speaking vestibular patients. J Vestib Res. 2016;25(5-6):253-9. doi: 10.3233/VES-160568. PMID 26890426
- [Result] Alghwiri AA, Khalil H, Al-Sharman A, El-Salem K. Psychometric properties of the Arabic Activities-specific Balance Confidence scale in people with multiple sclerosis: Reliability, validity, and minimal detectable change. NeuroRehabilitation. 2020;46(1):119-125. doi: 10.3233/NRE-192900. PMID 32039869
- [Result] Elboim-Gabyzon M, Agmon M, Azaiza F. Psychometric properties of the Arabic version of the Activities-Specific Balance Confidence (ABC) scale in ambulatory, community-dwelling, elderly people. Clin Interv Aging. 2019 Jun 18;14:1075-1084. doi: 10.2147/CIA.S194777. eCollection 2019. PMID 31354251
- [Result] Burger H, Giordano A, Bavec A, Franchignoni F. The Prosthetic Mobility Questionnaire, a tool for assessing mobility in people with lower-limb amputation: validation of PMQ 2.0 in Slovenia. Int J Rehabil Res. 2019 Sep;42(3):263-269. doi: 10.1097/MRR.0000000000000354. PMID 31210649